CLINICAL TRIAL: NCT01343264
Title: Trimodality Therapy for Malignant Pleural Mesothelioma: Radical Pleurectomy, Followed by Adjuvant Chemotherapy With Cisplatin/Pemetrexed and Radiotherapy
Brief Title: Trimodality Therapy for Malignant Pleural Mesothelioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HSK Wiesbaden (Other)
Responsible Party: Prof. Dr. Joachim Schirren, HSK Wiesbaden
Other Study IDs: RP2002-01
Record Dates: First submitted 2011-04-05; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Radical Pleurectomy; Pleurectomy/decortication; Cisplatin; Pemetrexed; Radiation
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The role of surgical resection in the management of Malignant Pleural Mesothelioma (MPM) is still controversial. The selection criterion to perform either Extrapleural Pneumonectomy (EPP) or Pleurectomy/Decortication (P/D) is dependent not only on the cardio-pulmonary status of the patient, tumor stage and intraoperative findings but also on surgeons' decision and philosophy. There are no established guidelines. Radical Pleurectomy (RP) competes against EPP as surgical therapy modality. Both surgical approaches are cytoreductive treatment options. The aim is to remove all gross disease and to achieve macroscopic complete resection.

Originally P/D was a palliative option for controlling pleural effusion. But lung-sparing surgery for MPM seems to be an alternative to patients unsuitable or unwilling to undergo EPP in a multimodality therapy concept. Most studies evaluating multimodality therapies for MPM are based on retrospective analyses and their interpretation is difficult because of inhomogeneous patient groups studied.

The aim of our study was to analyze the feasibility and results of RP as surgical therapy modality in a standardized trimodality therapy concept.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of MPM (all subtypes)
* Clinical T1-3, N0-2, M0 disease.
* No prior treatment for MPM.
* Adequate renal and liver function
* Adequate cardio-pulmonary reserves

Exclusion Criteria:

* Patients with unresectable disease
* Patients with an active infection that require systemic treatments
* Patients with a concurrent active malignancy.
* Patients with serious medical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant pleural mesothelioma prsentint at the Deparment of Thoracic Surgery, HSK Wiesbaden
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-11; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine the overall 5-year survival rate. | 5-years

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months
  Morbidity
Number of Participants with treatment related deaths as a Measure of Safety and Tolerability | 3 months
  Mortality
Recurrence | 5 years
  Occurence of tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schirren, MD, PhD, Principal Investigator — HSK Wiesbaden
Locations (1):
- Dr. Horst Schmidt Klinik, Department of Thoracic Surgery, Wiesbaden, Germany